CLINICAL TRIAL: NCT04384523
Title: A Phase 1 Randomized, Double Blinded, Placebo-Controlled Single Dose Escalation Study of OsrHSA in Adult Healthy Male and Female Volunteers
Brief Title: A Study of OsrHSA in Adult Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Healthgen Biotechnology Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: US-HY1001
Record Dates: First submitted 2020-04-13; First posted 2020-05-12 (Actual); Results first posted 2021-06-01 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Ascites Hepatic
Keywords: OsrHSA

STUDY DESIGN:
Intervention Model Description: This is a Phase 1 randomized, double blinded, placebo-controlled, single dose escalation study in healthy volunteers to evaluate safety, tolerability, PK, PD and immunogenicity of OsrHSA.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- OsrHSA 20 mg/kg IV (Experimental)
  Interventions: Drug: OsrHSA 20 mg/kg IV; Other: Placebo
- OsrHSA 40 mg/kg IV (Experimental)
  Interventions: Drug: OsrHSA 40 mg/kg IV; Other: Placebo
- OsrHSA 80 mg/kg IV (Experimental)
  Interventions: Drug: OsrHSA 80 mg/kg IV; Other: Placebo
- OsrHSA 140 mg/kg IV (Experimental)
  Interventions: Drug: OsrHSA 140 mg/kg IV; Other: Placebo
- OsrHSA 200 mg/kg IV (Experimental)
  Interventions: Drug: OsrHSA 200 mg/kg IV; Other: Placebo

INTERVENTIONS:
Drug: OsrHSA 20 mg/kg IV — A single dose of OsrHSA 20 mg/kg IV infusion at a rate lower than 2 ml/min
  Arms: OsrHSA 20 mg/kg IV
Drug: OsrHSA 40 mg/kg IV — A single dose of OsrHSA 40 mg/kg IV infusion at a rate lower than 2 ml/min
  Arms: OsrHSA 40 mg/kg IV
Drug: OsrHSA 80 mg/kg IV — A single dose of OsrHSA 80 mg/kg IV infusion at a rate lower than 2 ml/min
  Arms: OsrHSA 80 mg/kg IV
Drug: OsrHSA 140 mg/kg IV — A single dose of OsrHSA 140 mg/kg IV infusion at a rate lower than 2 ml/min
  Arms: OsrHSA 140 mg/kg IV
Drug: OsrHSA 200 mg/kg IV — A single dose of OsrHSA 200 mg/kg IV infusion at a rate lower than 2 ml/min
  Arms: OsrHSA 200 mg/kg IV
Other: Placebo — Normal Saline (0.9% Sodium Chloride)

SUMMARY:
A Phase 1 randomized, double blinded, placebo-controlled single dose escalation study of OsrHSA in adult healthy male and female volunteers

DETAILED DESCRIPTION:
This is a Phase 1 randomized, double blinded, placebo-controlled, single dose escalation study to evaluate safety, tolerability, PK, and immunogenicity of OsrHSA in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the following criteria to be enrolled in the trial

1. Able to understand and willing to sign the ICF
2. Healthy male and female subjects, 18-55 years of age, non-smokers, or subjects must have been non-smoking for at least 3 months prior to their screening visit.
3. Has adequate venous access
4. With no significant medical history, and in good health as determined by detailed medical history (neurological, endocrinal, cardiovascular, pulmonary, hematological, immunologic, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease), full physical examination,vital signs, 12-lead electrocardiogram (ECG), urinalysis and laboratory tests at screening. For eligibility purposes, abnormal laboratory or vital signs results may be repeated once if abnormal result is observed at the initial reading. Moreover, abnormalities found in the ECG may need to be confirmed by repeated measurements.
5. Subjects must have adequate organ function according to the following laboratory values:

   * Bone marrow function (absolute neutrophil count ≥1500/mm3 and platelet count ≥100,000/mm3)
   * Adequate liver function [alanine aminotransferase (ALT) to ≤1.5× upper limit normal (ULN) and alkaline phosphatase to ≤1.5× ULN, total bilirubin ≤1.5 mg/dL]
   * Adequate renal function creatinine clearance ≥60 mL/min based on Cockcroft- Gault equation, or serum creatinine level ≤1.5 times the ULN.
6. Be a female of non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is 2 years post-menopausal and have an FSH > 40mIU/mL, or surgically sterile [defined as having a bilateral oophorectomy, hysterectomy or tubal ligation]) or agree to one of the following to prevent pregnancy and, if a woman of childbearing potential, have a negative urine pregnancy test at screening:

   * Practicing abstinence
   * If a sexually active woman of childbearing potential (sexually active with a non-sterile male partner) agrees to prevent pregnancy by using double methods of contraception as follow until at least 30 days after the administration of the investigational product:

     1. simultaneous use of intra-uterine contraceptive device, placed at least 4 weeks prior to study drug administration, and condom for the male partner;
     2. simultaneous use of hormonal contraceptives, starting at least 4 weeks prior to study drug administration and must agree to use the same hormonal contraceptive throughout the study, and condom for the male partner;
     3. simultaneous use of diaphragm with intravaginally applied spermicide and male condom for the male partner, starting at least 21 days prior to study drug administration.
   * Male subjects who are not vasectomized for at least 6 months and who are sexually active with a non-sterile female partner must agree to use double methods of contraception below from the first dose of randomized study drug until 90 days after their dose and must not donate sperm during their study participation period:

     1. Simultaneous use of a male condom and, for the female partner, hormonal contraceptives (used since at least 4 weeks) or intra-uterine contraceptive device (placed since at least 4 weeks);
     2. Simultaneous use of a male condom and, for the female partner, a diaphragm with intravaginally applied spermicide.
7. Body mass index (BMI) 18-30 kg/m2 and body weight ≥ 50.0 kg for males and ≥ 45.0 kg for females.
8. Blood pressure ≤ 139/89 mm Hg.
9. Subjects are able to follow the study protocol and complete the trial.
10. At least 25% of the enrolled subjects will be of Asian descent, defined as Chinese, Japanese, Korean, Vietnamese, Hmong, and their offspring.

Exclusion Criteria:

Subjects who meet any of the following criteria cannot be enrolled:

1. History of severe infection within 4 weeks to dosing.
2. Signs and symptoms of any active infection regardless of severity within 2 weeks prior to dosing.
3. Meals & Dietary Restrictions: No seafood or high-fat food will be served during confinement in the clinical center
4. Subjects who have any history of allergy to food or drug will be excluded ( Including allergies, hypersensitivity, or intolerance to rice or rice products )
5. Use of any prescription drugs, herbal supplements, or nonprescription drugs including oral anti-histamines (for seasonal allergies) within 1 month or 5 half-lives (whichever is longer) prior to study drug administration, or dietary supplements within 1 week prior to study drug administration, unless, in the opinion of the Investigator and Sponsor, the medication will not interfere with the study. Over-the-counter multivitamins will be permitted. If needed, paracetamol/acetaminophen may be used, but must be documented in the Concomitant medications/Significant non-drug therapies page of the source data. Any questions of concomitant medications should be directed to the Sponsor.
6. Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to the first dosing, administration of a biological product in the context of a clinical research study within 90 days prior to the first dosing, or concomitant participation in an investigational study involving no drug or device administration.
7. Donation of blood 12 week prior to dosing.
8. Pregnant, or nursing females.
9. A history of substance abuse, psychiatric and psychological condition that, in the judgment of the investigator, may interfere with the planned treatment and follow-up, affect subject compliance or place the subject at high risk from treatment-related complications
10. A history of severe allergic reaction to any HpHSA component.
11. A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTcF interval >450 milliseconds [ms])
12. History of or active obstructive disease in biliary tract, liver, kidney and spleen defined by ultrasound.
13. Subjects who test positive for hepatitis B or C. (no matter carriers or active will be excluded from the study
14. Subjects who test positive for Syphilis, Human immunodeficiency virus (HIV) positive will also be excluded from the study.
15. Immunization with a live or attenuated vaccine is prohibited within 4 weeks prior to study drug administration. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed)
16. Positive Ig E and Ig G against rice at screening
17. History of significant alcohol abuse within one year prior to screening or regular use of alcohol within six months prior to the screening visit (more than fourteen units of alcohol per week [1 unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol]) or positive alcohol breath test at screening
18. History of significant drug abuse within one year prior to screening or use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine [PCP], crack, opioid derivatives including heroin, and amphetamine derivatives) within 1 year prior to screening
19. Positive urine drug screen, cotinine test, or alcohol breath test at screening
20. Any reason which, in the opinion of the Qualified Investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Nguyen, MD, MBA, Principal Investigator — WCCT Global, Inc
Locations (1):
- WCCT Global, Inc, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | OsrHSA 20 mg/kg IV | OsrHSA 40 mg/kg IV | OsrHSA 80 mg/kg IV | OsrHSA 140 mg/kg IV | OsrHSA 200 mg/kg IV
Started | 10 | 6 | 6 | 6 | 7 | 6
Completed | 9 | 5 | 6 | 6 | 7 | 5
Not Completed | 1 | 1 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | OsrHSA 20 mg/kg IV | OsrHSA 40 mg/kg IV | OsrHSA 80 mg/kg IV | OsrHSA 140 mg/kg IV | OsrHSA 200 mg/kg IV | Total
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 7 | 6 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.1 (8.82) | 34.2 (6.15) | 33.0 (7.13) | 35.3 (10.67) | 37.1 (9.49) | 36.0 (2.28) | 35.4 (7.67)
Age, Continuous [Median (Full Range); unit: years] | 33.0 [22 to 50] | 34.5 [26 to 44] | 33.5 [25 to 41] | 34.0 [22 to 54] | 37.0 [22 to 50] | 35.5 [34 to 40] | 35.0 [22 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 4 | 1 | 5 | 4 | 23
  Male | 5 | 2 | 2 | 5 | 2 | 2 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3 | 1 | 0 | 2 | 9
  Not Hispanic or Latino | 10 | 3 | 3 | 5 | 7 | 4 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 3 | 0 | 1 | 1 | 3 | 2 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 1 | 2 | 2 | 1 | 11
  White | 4 | 3 | 4 | 3 | 2 | 3 | 19
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: Kilograms] | 61.8 (10.78) | 67.6 (13.51) | 68.2 (4.35) | 72.2 (10.36) | 76.0 (23.21) | 68.7 (17.56) | 68.6 (14.40)
Weight [Median (Full Range); unit: Kilograms] | 62.5 [46.1 to 79.0] | 67.2 [45.9 to 87.3] | 69.4 [60.3 to 73.2] | 71.6 [57.5 to 86.1] | 83 [47.0 to 101.2] | 68.1 [49.0 to 88.4] | 67.3 [45.9 to 101.2]
Height [Mean (Standard Deviation); unit: Centimeter] | 167.3 (8.59) | 165.7 (12.15) | 162.8 (8.47) | 173.4 (8.06) | 170.9 (12.22) | 168.3 (14.06) | 168.1 (10.49)
Height [Median (Full Range); unit: Centimeter] | 167.5 [155.6 to 178.3] | 169.0 [148.1 to 179.9] | 161.4 [155.2 to 177.6] | 171.8 [163.6 to 187.3] | 171.1 [155.4 to 186.3] | 165.8 [154.0 to 192.9] | 169.1 [148.1 to 192.9]
BMI [Mean (Standard Deviation); unit: kg/m2] | 22.0 (3.16) | 24.4 (2.91) | 25.8 (2.46) | 24.0 (2.50) | 25.4 (4.58) | 23.9 (3.32) | 24.1 (3.35)
BMI [Median (Full Range); unit: kg/m2] | 21.4 [17.8 to 29.3] | 23.6 [20.9 to 28.8] | 25.8 [21.8 to 29.0] | 24.8 [19.7 to 26.5] | 28.4 [19.5 to 29.3] | 22.8 [20.7 to 28.6] | 23.6 [17.8 to 29.3]

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-Emergent Adverse Events
Time Frame: from date of Informed Consent through Day 30 (Study Completion)
Measure: Count of Participants; unit: Participants
Groups:
- OsrHSA 20 mg/kg IV: A single dose of OsrHSA 20 mg/kg IV
- OsrHSA 40 mg/kg IV: A single dose of OsrHSA 40 mg/kg IV
- OsrHSA 80 mg/kg IV: A single dose of OsrHSA 80 mg/kg IV
- OsrHSA 140 mg/kg IV: A single dose of OsrHSA 140 mg/kg IV
- OsrHSA 200 mg/kg IV: A single dose of OsrHSA 200 mg/kg IV
Arm/Group | Placebo | OsrHSA 20 mg/kg IV | OsrHSA 40 mg/kg IV | OsrHSA 80 mg/kg IV | OsrHSA 140 mg/kg IV | OsrHSA 200 mg/kg IV
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 7 | 6
Participants | 1 | 0 | 2 | 1 | 2 | 0

2. Secondary Outcome: Maximum Plasma Concentration [Cmax]
Time Frame: pre-dose, 0.5 hours after dose initiating, EOI (End of Infusion), and 0.5 hours, 4 hours, 12 hours, 24 hours (Day 2), 48 hours (Day 3), Day 5, Day 8, Day 15, Day 22, and Day 30 post End of Infusion.
Reporting Status: Not Posted

3. Secondary Outcome: Number of Participants With ADA Incident Events
Time Frame: pre-dose, Day 8, Day 15, Day 22, and Day 30 post End of Infusion
Measure: Number; unit: participants
Arm/Group | Placebo | OsrHSA 20 mg/kg IV | OsrHSA 40 mg/kg IV | OsrHSA 80 mg/kg IV | OsrHSA 140 mg/kg IV | OsrHSA 200 mg/kg IV
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 7 | 6
participants | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Screening to Day 30 +/- 2 days
Arm/Group | Placebo | OsrHSA 20 mg/kg IV | OsrHSA 40 mg/kg IV | OsrHSA 80 mg/kg IV | OsrHSA 140 mg/kg IV | OsrHSA 200 mg/kg IV
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6 | 0/6 | 0/6 | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/6 | 0/6 | 0/6 | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 1/10 | 0/6 | 2/6 | 1/6 | 2/7 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | OsrHSA 20 mg/kg IV (N=6) | OsrHSA 40 mg/kg IV (N=6) | OsrHSA 80 mg/kg IV (N=6) | OsrHSA 140 mg/kg IV (N=7) | OsrHSA 200 mg/kg IV (N=6)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-11-20): https://cdn.clinicaltrials.gov/large-docs/23/NCT04384523/Prot_SAP_001.pdf
  • Informed Consent Form (2019-11-14): https://cdn.clinicaltrials.gov/large-docs/23/NCT04384523/ICF_000.pdf